CLINICAL TRIAL: NCT04879602
Title: Second Affiliated Hospital of Zhejiang University,School of Medicine
Brief Title: Effect of Suctioning by Bronchoscope on Postoperative Pulmonary Complications Among Patients With SCI in the PACU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0162
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Suction; Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchoscopy group (Experimental): patients receive suction before extubation by bronchoscopy in PACU
  Interventions: Behavioral: suction with bronchoscopy
- Control group (No Intervention): patients receive routine ordinary suction in PACU

INTERVENTIONS:
Behavioral: suction with bronchoscopy — suction with bronchoscopy
  Arms: Bronchoscopy group

SUMMARY:
Respiratory failure and dyspnea are common in spinal cord injury (SCI), and in acute situations, any spinal cord lesion above T11 can cause abnormal respiratory function and impair the airway clearance.

Although surgical decompression is one of the key early neuroprotective therapies, surgery and general anesthesia disrupt many aspects of respiratory function and may cause a series of postoperative pulmonary complications.

Endotracheal suction is important to reduce the risk of lung consolidation and atelectasis. But for patients with respiratory insufficiency such as SCI, ordinary suction is not enough to clear secretions in the deeper airways. And repeated intratracheal suction may even cause some serious complications.

Bronchoscopy can generally penetrate into the bronchus of grade 3-4, and fully attract the secretions in it under visual conditions. Its curative effect on pneumonia and atelectasis in the ICU has been affirmed, but no one has yet explored the application in the postoperative care unit .

DETAILED DESCRIPTION:
All patients admitted to PACU with tracheal tube after operation will be recruited, and than be randomly divided into two groups during resuscitation:

1. one group receives routine ordinary sputum suction ; the other group receives routine ordinary sputum suction with bronchoscopy
2. After entering the PACU, both groups will receive two lung ultrasound examinations and record the lung ultrasound scores: when entering PACU and when leaving PACU.

After returning to the ward, the doctor in charge will make medical decisions and treatments based on the condition.

Follow up for pulmonary complications (respiratory tract infection, respiratory failure, bronchospasm, atelectasis, pleural effusion, pneumothorax, pulmonary edema, pulmonary embolism, aspiration pneumonia) within 7 days after surgery.

Follow-up 30 days and 90 days after operation.

ELIGIBILITY:
Inclusion Criteria:

- Age>=18 Spinal injury level :above T11 Stable preoperative spontaneous respiration Elective cervical/thoracic spine fixation American Spinal Injury Association (ASIA) class: A-D

Exclusion Criteria:

- Unconscious before surgery Pregnant With mental disorders Directly transfered to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative pulmonary complications | within 7 days after operation or before discharge, whichever came first
  postoperative pulmonary complications are defined as a composite outcome including respiratory infection, respiratory failure,pleural effusion, atelectasis,pneumothorax,broncospasm and aspiration pneumonitis postoperative pulmonary complications are defined as a composite outcome including respiratory infection, respiratory failure,pleural effusion, atelectasis,pneumothorax,broncospasm and aspiration pneumonitis
  including respiratory infection, respiratory failure,pleural effusion, atelectasis, pneumothorax , broncospasm and aspiration pneumonitis

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, MD, Study Chair — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No